CLINICAL TRIAL: NCT02060539
Title: Multicenter Dispensing Study of Biofinity Lenses in Extended Range
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-13-47
Record Dates: First submitted 2014-02-06; First posted 2014-02-12 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2015-06

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biofinity XR (Experimental): Participants dispensed Biofinity XR lenses over two weeks of lens wear
  Interventions: Device: Biofinity XR

INTERVENTIONS:
Device: Biofinity XR

SUMMARY:
To obtain subjective and objective feedback on the clinical performance of Biofinity lenses after at least two weeks daily wear in existing contact lens wearers compared with their habitual lenses.

ELIGIBILITY:
Inclusion Criteria:

* Has had an oculo-visual examination in the last two years
* Is at least 18 years of age and has full legal capacity to volunteer
* Has read and understood the information consent letter
* Is willing and able to follow instructions and maintain the appointment schedule
* Is correctable to a visual acuity of 20/50 or better (in at least one eye) with their habitual vision correction
* Currently wears soft contact lenses
* They should require contact lens powers between -12.00 and -20.00D or between +8.00 and +15.00D
* Has clear corneas and no active ocular disease
* Demonstrates an acceptable fit with the study lenses.

Exclusion Criteria:

* Has any systemic disease affecting ocular health
* Is taking medication, such as antihistamine eye drops, oral and ophthalmic betaadrenergic blockers (e.g. Propanolol, Timolol), anticholinergics, and any prescribed or over-the-counter eye medication, except artificial tears or eye lubricants
* Have any active ocular disease and/or infection that would contraindicate contact lens wear.
* Active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.
* Has worn gas permeable contact lenses within the last month.
* Is aphakic
* Has undergone corneal refractive surgery.
* Is participating in any other type of clinical research study
* Female who is currently pregnant or is breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, Principal Investigator — CCLR, University of Waterloo; Meng Lin, Principal Investigator — CRC, University of California Berkeley; Jan Bergmanson, Principal Investigator — TERTC, University of Houston; Pete Kollbaum, Principal Investigator — CORL, Indiana University
Locations (4):
- United States (3):
  - UC Berkeley Clinica Research Center, Berkeley, California
  - CORL, Indiana University School of Optometry, Indianapolis, Indiana
  - TERTC, University of Houston, Houston, Texas
- CCLR, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study included 2 visits screening and fitting. Up to 50 existing lens wearers prescriptions from +20 to -20D spheres fitted. Participants evaluated at baseline/screening and lens dispensing visit with at least 1 other visit occurring at minium of 2 weeks lens wear.
Groups:
- Comfilcon A: Participants dispensed Biofinity XR lenses over two weeks of lens wear
  Biofinity XR / comfilcon A
Period: Overall Study
Arm/Group | Comfilcon A
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Region of Enrollment [Number; unit: participants]
  Canada | 4
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Dryness (During Day and Dryness at Night)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=cannot be worn, Extremely dry. 100=No dryness experienced at any time.) Obtained habitual lens history at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale
  Dryness During Day | 69 (17)
  Dryness at End of Day | 53 (25)

2. Secondary Outcome: Lens Centration - Habitual Lenses
Description: Objective measurement by investigator. (Assessed as optimum, slightly decentered, extremely decentered) Obtained for habitual lenses at baseline.
Time Frame: Baseline
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Lenses) | 38
percentage of lenses
  optimum | 53
  slightly decentered | 37
  extremely decentered | 11

3. Primary Outcome: Dryness (During Day)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=cannot be worn, Extremely dry. 100=No dryness experienced at any time.) Obtained at dispense; Lens pair one dispensed at the baseline visit and Lens pair two dispensed at 2 weeks visit.
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 92 (10)

4. Primary Outcome: Dryness (During Day and Dryness at Night)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=cannot be worn, Extremely dry. 100=No dryness experienced at any time.) Obtained at two weeks.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale
  Dryness | 87 (12)
  Dryness at End of Day | 76 (24)

5. Primary Outcome: Comfort (Insertion, End of Day, Overall)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=cannot be worn,Causes pain; 100=Cannot be felt ever) Obtained habitual lens history at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale
  Comfort | 86 (8)
  Comfort at End of Day | 62 (18)
  Overall Comfort | 83 (15)

6. Primary Outcome: Comfort (Insertion)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=cannot be worn,Causes pain; 100=Cannot be felt ever) Obtained at dispense; Lens pair one dispensed at the baseline visit and Lens pair two dispensed at 2 weeks visit.
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 89 (9)

7. Primary Outcome: Comfort (Insertion, End of Day, Overall)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=cannot be worn,Causes pain; 100=Cannot be felt ever) Obtained at 2 weeks.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale
  Comfort | 89 (11)
  Comfort at End of Day | 76 (22)
  Overall Comfort | 86 (17)

8. Primary Outcome: Ghosting (Multiple Images)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extreame ghosting. Cannot be worn. 100=No ghosting ever.) Obtained habitual lens history at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 90 (12)

9. Primary Outcome: Ghosting (Multiple Images)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extreme ghosting. Cannot be worn. 100=No ghosting ever.) Obtained at dispense; Lens pair one dispensed at the baseline visit and Lens pair two dispensed at 2 weeks visit.
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 93 (15)

10. Primary Outcome: Ghosting (Multiple Images)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extreme ghosting. Cannot be worn. 100=No ghosting ever.) Obtained at 2 weeks.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 92 (15)

11. Primary Outcome: Hazing (Blurred Edges)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extreame haze. Cannot be worn. 100=No hazing experienced at any time.) Obtained habitual lens history at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 79 (24)

12. Primary Outcome: Hazing (Blurred Edges)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extreme haze. Cannot be worn. 100=No hazing experienced at any time.) Obtained at 2 weeks.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 92 (14)

13. Primary Outcome: Vision Quality (During Day and at Night)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extremely poor vision all the time. Cannot function; 100=Excellent vision all of the time.) Obtained habitual lens history at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale
  Vision During the Day | 78 (17)
  Vision at Night | 62 (22)

14. Primary Outcome: Vision Quality (During Day)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extremely poor vision all the time. Cannot function; 100=Excellent vision all of the time.) Obtained at dispense; Lens pair one dispensed at the baseline visit and Lens pair two dispensed at 2 weeks visit.
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 87 (15)

15. Primary Outcome: Vision Quality (During Day and at Night)
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extremely poor vision all the time. Cannot function; 100=Excellent vision all of the time.) Obtained at 2 weeks.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale
  Vision During the Day | 86 (16)
  Vision at Night | 78 (22)

16. Primary Outcome: Handling (Insertion, Removal, Overall)
Description: as for outcome 5
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale
  Ease of Insertion | 93 (10)
  Ease of Removal | 87 (13)
  Ease of Handling Overall | 91 (12)

17. Primary Outcome: Handling (Insertion, Removal, Overall)
Description: as for outcome 7
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale
  Ease of Insertion | 94 (7)
  Ease of Removal | 83 (19)
  Ease of Handling Overall | 89 (13)

18. Primary Outcome: Overall Satisfaction of Comfort, Vision, Handling
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extremely dissatisfied; 100=Extremely satisfied.) Obtained at dispense; Lens pair one dispensed at the baseline visit and Lens pair two dispensed at 2 weeks visit.
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 90 (8)

19. Primary Outcome: Overall Satisfaction of Comfort, Vision, Handling
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extremely dissatisfied; 100=Extremely satisfied.) Obtained habitual lens history at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 82 (15)

20. Primary Outcome: Overall Satisfaction of Comfort, Vision, Handling
Description: Subjective response of participant by questionnaire on a visual analog scale (0-100, 0=Extremely dissatisfied; 100=Extremely satisfied.) Obtained at baseline at 2 weeks.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
units on a scale | 87 (15)

21. Primary Outcome: Comfort Preference
Description: Subjective response of participant by questionnaire on a likert scale (Prefer New Lenses Strongly, Prefer New Lenses Slightly, No Preference - both acceptable/both unacceptable, Prefer My Own Lenses Slightly, Prefer My Own Lenses Strongly) Obtained at dispense; Lens pair one dispensed at the baseline visit and Lens pair two dispensed at 2 weeks visit.
Time Frame: Dispense
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
percentage of participants
  comfilcon A lenses | 47
  habitual lenses | 16
  no preference | 37

22. Primary Outcome: Comfort Preference
Description: Subjective response of participant by questionnaire on a likert scale (Prefer New Lenses Strongly, Prefer New Lenses Slightly, No Preference - both acceptable/both unacceptable, Prefer My Own Lenses Slightly, Prefer My Own Lenses Strongly) Obtained at 2 weeks.
Time Frame: 2 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
percentage of participants
  comfilcon A lenses | 42
  habitual lenses | 26
  no preference | 32

23. Primary Outcome: Vision Preference
Description: as for outcome 21
Time Frame: Dispense
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
percentage of participants
  comfilcon A lenses | 42
  habitual lenses | 0
  no preference | 58

24. Primary Outcome: Vision Preference
Description: as for outcome 22
Time Frame: 2 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
percentage of participants
  comfilcon A lenses | 53
  habitual lenses | 31
  no preference | 16

25. Primary Outcome: Handling Preference
Description: as for outcome 22
Time Frame: 2 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
percentage of participants
  comfilcon A lenses | 32
  habitual lenses | 32
  no preference | 37

26. Primary Outcome: Overall Preference
Description: as for outcome 21
Time Frame: Dispense
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
percentage of participants
  comfilcon A lenses | 37
  habitual lenses | 5
  no preference | 58

27. Primary Outcome: Overall Preference
Description: as for outcome 22
Time Frame: 2 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
percentage of participants
  comfilcon A lenses | 63
  habitual lenses | 21
  no preference | 16

28. Secondary Outcome: Lens Centration
Description: Objective measurement by investigator. (Assessed as optimum, slightly decentered, extremely decentered) Obtained at baseline at dispense.
Time Frame: Dispense
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Lenses) | 38
percentage of lenses
  optimum | 63
  slightly decentered | 26
  extremely decentered | 10

29. Secondary Outcome: Lens Centration
Description: Objective measurement by investigator. (Assessed as optimum, slightly decentered, extremely decentered) Obtained at 2 weeks.
Time Frame: 2 Weeks
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Lenses) | 38
percentage of lenses
  optimum | 63
  slightly decentered | 32
  extremely decentered | 5

30. Secondary Outcome: Lens Movement - Habitual Lenses
Description: Objective measurement by investigator of overall post-blink lens movement. (Average Grade; Graded 0-4; 0=exceptionally tight, 2=optimal, 4=exceptionally loose) Obtained for habitual lenses at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Lenses) | 38
units on a scale | 2.47 (0.92)

31. Secondary Outcome: Lens Movement
Description: Objective measurement by investigator of overall post-blink lens movement. (Average Grade; Graded 0-4; 0=exceptionally tight, 2=optimal, 4=exceptionally loose) Obtained at dispense; Lens pair one dispensed at the baseline visit and Lens pair two dispensed at 2 weeks visit.
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Lenses) | 38
units on a scale | 2.39 (0.52)

32. Secondary Outcome: Lens Movement
Description: Objective measurement by investigator of overall post-blink lens movement. (Average Grade; Graded 0-4; 0=exceptionally tight, 2=optimal, 4=exceptionally loose) Obtained at 2 weeks wear.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Lenses) | 38
units on a scale | 2.45 (0.60)

33. Secondary Outcome: Overall Fit Acceptance
Description: Objective measurement by investigator of overall fit acceptance. (scale 0-4; 0=very poor, 4=very good) Obtained for habitual lenses at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Lenses) | 38
units on a scale | 3.33 (0.59)

34. Secondary Outcome: Overall Fit Acceptance
Description: Objective measurement by investigator of overall fit acceptance. (scale 0-4; 0=very poor, 4=very good) Obtained at dispense; Lens pair one dispensed at the baseline visit and Lens pair two dispensed at 2 weeks visit.
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Lenses) | 38
units on a scale | 3.47 (0.51)

35. Secondary Outcome: Overall Fit Acceptance
Description: Objective measurement by investigator of overall fit acceptance. (scale 0-4; 0=very poor, 4=very good) Obtained at 2 weeks.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Lenses) | 38
units on a scale | 3.45 (0.394)

36. Secondary Outcome: Visual Acuity
Description: Objective measurement by investigator of monocular high and low contrast logMar visual acuity. Visual Acuity High-Contrast (VA HC), Visual Acuity Low-Contrast (VA LC), Visual Acuity High-Contrast OU (VA HC OU), Visual Acuity Low-Contrast OU (VA LC OU). Obtained for habitual lenses at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: logMar
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
logMar
  VA HC | 0.16 (0.12)
  VA LC | 0.22 (0.14)
  VA HC (OU) | 0.04 (0.13)
  VA LC (OU) | 0.15 (0.15)

37. Secondary Outcome: Visual Acuity
Description: Objective measurement by investigator of monocular high and low contrast logMar visual acuity. Visual Acuity High-Contrast (VA HC), Visual Acuity Low-Contrast (VA LC), Visual Acuity High-Contrast OU (VA HC OU), Visual Acuity Low-Contrast OU (VA LC OU). Obtained at dispense; Lens pair one dispensed at the baseline visit and Lens pair two dispensed at 2 weeks visit.
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: logMar
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
logMar
  VA HC | 0.10 (0.15)
  VA LC | 0.18 (0.16)
  VA HC (OU) | 0.03 (0.13)
  VA LC (OU) | 0.11 (0.14)

38. Secondary Outcome: Visual Acuity
Description: Objective measurement by investigator of monocular high and low contrast logMar visual acuity. Visual Acuity High-Contrast (VA HC), Visual Acuity Low-Contrast (VA LC), Visual Acuity High-Contrast OU (VA HC OU), Visual Acuity Low-Contrast OU (VA LC OU). Obtained at 2 weeks.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: logMar
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
logMar
  VA HC | 0.11 (0.11)
  VA LC | 0.18 (0.15)
  VA HC (OU) | 0.02 (0.12)
  VA LC (OU) | 0.11 (0.14)

39. Secondary Outcome: Anterior Ocular Physiological Response
Description: Ocular response assessed with the slit lamp using a Visual Analog Scale (0-4, 0=none, 4=severe). Obtained for habitual lenses at baseline.
Time Frame: Baseline
Population: Overall Conjunctival Staining (n=16), Overall Palpebral Papillae (n=8) Missing data as not all sites collected this data.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Eyes) | 38
units on a scale
  Overall Redness Bulbar | 1.13 (0.64)
  Overall Redness Limbal | 0.84 (0.78)
  Overall Corneal Staining Type | 0.68 (0.53)
  Corneal Staining Extent (n=19) | 0.66 (0.58)
  Conjunctival Staining (n=16) | 0.31 (0.55)
  Overall Palpebral Injection | 0.8 (0.69)
  Overall Palpebral Papillae (n=8) | 0.3 (0.51)

40. Secondary Outcome: Anterior Ocular Physiological Response
Description: Ocular response assessed with the slit lamp using a Visual Analog Scale (0-4, 0=none, 4=severe). Obtained at 2 weeks.
Time Frame: 2 Weeks
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
Number analyzed (Eyes) | 38
units on a scale
  Overall Redness Bulbar | 1.00 (0.69)
  Overall Redness Limbal | 0.74 (0.81)
  Overall Corneal Staining Type | 0.47 (0.61)
  Corneal Staining Extent (n=19) | 0.45 (0.60)
  Conjunctival Staining (n=16) | 0.94 (0.96)
  Overall Palpebral Injection | 0.9 (0.61)
  Overall Palpebral Papillae (n=8) | 0.7 (0.65)

41. Secondary Outcome: Average Wearing Time
Description: Participant response when asked, "Number of hours worn today?" (hours per day) Obtained for habitual lens at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
hours | 13 (3.6)

42. Secondary Outcome: Average Wearing Time
Description: Participant response when asked, "Number of hours worn today?" (hours per day) Obtained at 2 weeks.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Comfilcon A
Number analyzed (Participants) | 19
hours | 12.5 (2.8)

ADVERSE EVENTS:
Arm/Group | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information gathered during this study is proprietary and should be made available only to those directly involved in the study. Information and reports arising from this project are the property of the sponsor.